CLINICAL TRIAL: NCT06941441
Title: Remotely-Monitored Exercise to Enhance Functional Outcomes in Patients With Pulmonary Arterial Hypertension (PAH) Initiating Sotatercept Therapy: A Single-site Feasibility Study
Brief Title: PAH Exercise Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Mary Beth Brown, Associate Professor, Department of Rehabilitation Medicine, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00021808
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Exercise Therapy
Keywords: PAH; pulmonary arterial hypertension; sotatercept; exercise
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise Arm (Experimental): Patients with PAH on sotatercept plus a tailored, progressive home exercise program with wrist-worn fitness tracker and oxygen saturation monitoring
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Home exercise program — A tailored, progressive home exercise program with wrist-worn fitness tracker and oxygen saturation monitoring

SUMMARY:
Ten patients with PAH who are stable and eligible to initiate sotatercept therapy will participate in a 26 week study that consists of a 24-week intervention period where patients will receive complimentary sotatercept as prescribed, plus a tailored, progressive home exercise program with wrist-worn fitness tracker and oxygen saturation monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented diagnostic right heart catheterization (RHC) at any time prior to screening confirming the diagnosis of WHO PAH Group 1 in any of the following subtypes: Idiopathic PAH, Heritable PAH, Drug/toxin-induced PAH, PAH associated with CTD, PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following repair
* Symptomatic PH classified as WHO FC II or III
* Baseline RHC performed during the Screening Period documenting a minimum PVR of ≥ 5 WU and a pulmonary capillary wedge (PCWP) or left ventricular end-diastolic pressure of ≤ 15 mmHg
* Receiving stable background therapy for PAH for >90 days and will continue receiving throughout trial. Background treatments may consist of monotherapy, double therapy, or triple therapy with currently available medications for PAH.
* Initiation of Sotatercept is clinically indicated
* Willing and able to participate in a remotely-monitored home exercise program for 24 weeks
* Ability to adhere to study visit schedule and understand and comply with all protocol requirements
* Ability to understand and provide written informed consent

Exclusion Criteria:

* Diagnosis of PH WHO Groups 2, 3, 4, or 5
* Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH, PAH associated with portal hypertension, schistosomiasis-associated PAH and pulmonary veno-occlusive disease
* Hemoglobin at screening above gender-specific ULN
* Baseline platelet count < 50,000/mm3 (< 50.0 × 109/L) at screening
* Uncontrolled systemic hypertension as evidenced by sitting systolic BP > 160 mmHg or sitting diastolic BP > 100 mmHg during screening visit after a period of rest; Baseline systolic BP < 90 mmHg at screening
* Pregnant or breastfeeding females
* Clinical laboratory liver and kidney function tests outside of normal range
* Currently enrolled in or have completed any other investigational product study within 30 days for small-molecule drugs or within 5 half-lives for biologics prior to the date of signed informed consent
* Prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536) or known allergic reaction to either one
* History of full pneumonectomy
* Initiation of a structured exercise program within 90 days prior or planned initiation during the study
* Known history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), defined as mild to severe hepatic impairment (Child-Pugh Class A-C).
* Cardiac related history: History of restrictive, constrictive, or congestive cardiomyopathy; History of atrial septostomy within 180 days prior to the screening visit; ECG with Fridericia's corrected QT interval (QTcF) > 500 ms during the Screening Period; Personal or family history of long QT syndrome (LQTS) or sudden cardiac death; Left ventricular ejection fraction (LVEF) < 45% on historical ECHO within 12 months prior to the screening visit; Any symptomatic coronary disease events (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain) within 6 months prior to the screening visit. Note: Anginal pain can be ignored as an exclusion criterion if coronary angiography shows no obstructions
* Cerebrovascular accident within 3 months prior to the screening visit
* Acutely decompensated heart failure within 14 days prior to the screening visit, as per investigator assessment
* Significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
* Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 18 months
Adherence and Completion Rate | 18 months
Study-related adverse events (SAE) rate | 18 months
Measurement fidelity for the innovative 'remote Six Minute Walk Test (6MWT)' | 18 months
  Patient self-administered via the digital fitness platform with remote monitoring at two interim assessment timepoints

SECONDARY OUTCOMES:
Change from baseline in Six Minute Walk Test (6MWT) distance | 24 weeks
  Via Six Minute Walk Test administered during baseline and final in-person study visits
Change from baseline in Calculated Cardiac Effort (CEC) during 6MWT | 24 weeks
  Cardiac Effort to be calculated from Six Minute Walk Test administered during baseline and final in-person study visits
Change from baseline in nT-proBNP | 24 weeks
  Via bloodwork during baseline and final in-person study visits
Average weekly accelerometry minutes of moderate-to-vigorous physical activity (MVPA) | 24 weeks
Health-related quality of life (QoL) | 24 weeks
  As measured by the PAH-specific survey PAH-SYMPACT®

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Brown, PT, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No